CLINICAL TRIAL: NCT03280290
Title: Partial Selective Depletion in Lymphocytes Transplant T CD4+ CCR7+ in Hematopoeitic Stem Cells Allograft
Brief Title: Transplant T CD4+ CCR7+ In Hematopoietic Stem Cells Allograft
Acronym: CCR7-CD4-DPL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010_09; 2010-A01231-38 (Other: ID-RDB number, ANSM)
Record Dates: First submitted 2014-06-24; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Acute Myeloblastic Leukemia
Keywords: Lymphocytes CD4; Lymphocytes CCR7; ALLOGRAFT; Hematopoietic Stem Cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- receivers (Experimental): * Eligible for allo-HSCs from peripheral blood stem cells from a compatible donor HLA family (Appendix 1, the pre-transplant assessment must be enabled)
  * In a complete remission rate of leucocytes with ≥ 2G / L
  * Affiliated to social security person or beneficiary of such a scheme.
  Interventions: Biological: blood
- Donors (Experimental): * Member of the siblings and HLA-matched A, B, Cw, DR, DQ
  * Eligible to donate peripheral blood stem cells for allo-HSCs (Appendix 2, pre donation assessment must be enabled)
  * Having a rate of circulating lymphocytes ≥ 1 G / L
  * Having a proportion of CD4 + CCR7 + ≥ 80% of the total CD4 T population
  * The statutes CMV and EBV are known (positive or negative).
  * Affiliated to social security person or beneficiary
  Interventions: Biological: blood

INTERVENTIONS:
Biological: blood — assessment pre-donation of hematopoietic stem cells (blood sample)

SUMMARY:
This is a preclinical study prior to the establishment of a cell therapy protocol applicable to humans.

The main objective is to evaluate the decrease in alloreactivity of TCD4 + population by partial selective depletion of CD4 + CCR7 + graft to less than 50 % of CD4 + totals. To test the alloreactivity of donor T lymphocytes.

DETAILED DESCRIPTION:
This is a preclinical study prior to the establishment of a cell therapy protocol applicable to humans.

The main objective is to evaluate the decrease in alloreactivity of TCD4 + population by partial selective depletion of CD4 + CCR7 + graft to less than 50 % of CD4 + totals. To test the alloreactivity of donor T lymphocytes , T lymphocytes CD4 + CCR7 + donor will be stimulated by mature dendritic cells (DC) derived from recipient circulating monocytes in a mixed lymphocyte reaction model sensitized ( MLDCR ) , experiencing HLA -compatibility . This first step will confirm the results previously obtained in a situation incompatible HLA .

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria of the receiver anti -infectious immunity

* Man or woman aged 18-65 years
* Eligible for allo - HSCs from peripheral blood stem cells from a compatible donor HLA family (Annex 3 , the pre- transplant assessment must be enabled)
* In a complete remission rate of leucocytes with ≥ 2G / L
* Affiliated to social security person or beneficiary of such a scheme.
* Having signed informed consent

Inclusion criteria for the study of the receiver of anti tumor immunity

* Man or woman aged 18-65 years
* Achieved a hyperleucocytic acute myelogenous leukemia ( leukocytes ≥ 20G / L)
* Patients whose blasts at diagnosis were cryopreserved in the tumor bank of the University Hospital of Lille (Professor Claude Prudhomme )
* Eligible for allo - HSCs from peripheral blood stem cells from a compatible donor HLA family (Annex 3 , the pre- transplant assessment must be enabled)
* In a complete remission rate of leucocytes with ≥ 2G / L
* Affiliated to social security person or beneficiary of such a scheme.
* Having signed informed consent receivers

Inclusion criteria of the donor

* Man or woman aged 18-65 years
* Member of the HLA-matched siblings and A, B, Cw, DR, DQ
* Eligible to donate peripheral blood stem cells for allo-HSCs (Appendix 2, pre donation assessment must be enabled)
* Having a rate of circulating lymphocytes ≥ 1 G / L
* Having a proportion of CD4 + CCR7 + ≥ 80% of the total CD4 T population
* The statutes CMV and EBV are known (positive or negative).
* Affiliated to social security person or beneficiary of such a scheme. who signed informed consent -

Exclusion Criteria:

Criteria for non inclusion of the pairs donor / Receiver

* Private person of liberty by judicial or administrative decision
* Person subject to a measure of legal protection
* Pregnant or breastfeeding woman
* People do not understand French or understanding with a disability.
* Major Protected Person in emergency and refusing or unable to give informed consent At any time, individuals may request to be removed from the study Each subject may come out of the study by decision of the competent administrative authority of the promoter and the coordinating investigator but also by decision of a co-investigator or by decision of the interested himself in accordance with regulations and as mentioned in the form of obtaining consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03-20 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change the lymphocyte proliferation will be evaluated using a scintillation spectrometer | 1 day, 5 day ,8 day
  Decrease in alloreactivity of TCD4.(composite) Decrease population by partial selective depletion of CD4 + CCR7 + graft to less than 50% of total CD4 +will be evaluated on this basis criteria.
Change the functional properties of cells will be evaluated by T-SPOT TB®. | 1 day, 5 day ,8 day
  Decrease in alloreactivity of TCD4.(composite) Decrease population by partial selective depletion of CD4 + CCR7 + graft to less than 50% of total CD4 +will be evaluated on this basis criteria.

SECONDARY OUTCOMES:
Response to anti-infectious immunity | 24 months
  Measure the anti-infectious immunity during a partial selective depletion of TCD4 + CCR7 + (≤ 50%)
Response to anti-tumor immunity | 24 months
  Measure the anti-tumor immunity during a partial selective depletion of TCD4 + CCR7 + (≤ 50%)

CONTACTS AND LOCATIONS:
Overall Officials: YAKOUB-AGHA IBRAHIM, Professor, Study Director — CHRU de Lille
Locations (1):
- Diseases of Blood Service HURIEZ hospital CHRU de LILLE, Lille, France

IPD SHARING:
Plan to Share IPD: No